CLINICAL TRIAL: NCT05413044
Title: A Nationwide Post-Marketing Study on the Safety of Abatacept Treatment in Sweden Using the SRQ Register
Brief Title: A Post-marketing Study to Assess the Safety of Abatacept in Sweden Using the Swedish Rheumatology Quality Register (SRQ) Register
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-816
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
Keywords: Abatacept; Orencia; Malignancies; Long-term safety follow-up
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Abatacept Group: Participants with established RA or PsA and receiving abatacept.
- Non-targeted Disease Modifying Anti-rheumatic Drug (DMARD) Group: Participants with established RA or PsA and not previously treated with any targeted DMARDs and who start treatment with a non-targeted DMARD.
- Targeted DMARD Group: Participants with established RA or PsA and previously treated without abatacept who start treatment with targeted DMARDs.

SUMMARY:
The purpose of this study is to collect real-world data in order to estimate the frequency of overall malignancies, melanoma, basal cell carcinoma, and squamous cell carcinoma in participants with rheumatoid arthritis (RA) or psoriatic arthritis (PsA) enrolled in the SRQ Register in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA or PsA
* ≥18 years at index treatment initiation
* Participants starting treatment with:
* abatacept
* non-targeted DMARDs
* targeted DMARD

Exclusion Criteria:

- Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RA or PsA who began abatacept, a non-targeted DMARD, or a targeted DMARD enrolled in the SRQ Register between January 2007 and January 2021.
Sampling Method: Non-Probability Sample
Enrollment: 140706 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Overall Malignancies | 5 years
Incidence Rate of Melanoma | 5 years
Incidence Rate of Non-melanoma Skin Cancer | 5 years
Incidence Rate of Basal Cell Carcinoma | 5 years
Incidence Rate of Squamous Cell Carcinoma | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html